CLINICAL TRIAL: NCT04731025
Title: Prophylactic Treatment of Breast Implants With a Solution of Gentamicin, Vancomycin and Cefazolin Antibiotics for Women Undergoing Breast Reconstructive Surgery: a Randomized Controlled Trial (The BREAST-AB Trial)
Brief Title: Local Antibiotics for Breast Implants
Acronym: BREAST-AB
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Mikkel Herly (Other)
Collaborators: University of Copenhagen (Other); Herlev and Gentofte Hospital (Other); Zealand University Hospital (Other); Odense University Hospital (Other); Vejle Hospital (Other); Esbjerg Hospital - University Hospital of Southern Denmark (Other); Aarhus University Hospital (Other); Aalborg University Hospital (Other)
Responsible Party: Sponsor-Investigator, Mikkel Herly, MD, Ph.d., Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: BREAST-AB-01; 2020-002459-40 (EudraCT Number); 0058322 (Other Grant/Funding Number: Novo Nordisk Foundation); R-189- A4127 (Other Grant/Funding Number: Medicine Fund of the Danish Regions)
Record Dates: First submitted 2021-01-26; First posted 2021-01-29 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-07

CONDITIONS: Implant Complication; Implant Infection; Implant Site Infection; Implant Capsular Contracture; Implant Site Pocket Infection; Implant Expulsion; Antibiotic Side Effect
MeSH Terms: conditions — Implant Capsular Contracture | interventions — Gentamicins; Cefazolin; Vancomycin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The trial will be double-blind so that the patients, site investigators and data monitors will be blinded to the allocation. Only the designated nurses and the members of the trial coordinating unit (who provide the randomization number and treatment allocation) are not blinded to the allocation. The unblinded persons will not in any way be part of the treatment, clinical evaluation of outcomes or data assessment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Irrigation of implants with sterile isotonic saline (Placebo Comparator): The placebo solution will consist of 500 mL of sterile isotonic (9%) saline contained in a infusion bag.
  Interventions: Other: Placebo
- Irrigation of implants with a triple antibiotic solution (Experimental): The antibiotic solution will contain 1000 mg vancomycin, 80 mg gentamicin and 1000 mg cefazolin in 500 mL sterile isotonic (9%) saline
  Interventions: Drug: Gentamicin, Cefazolin and Vancomycin

INTERVENTIONS:
Drug: Gentamicin, Cefazolin and Vancomycin — The antibiotic solution will contain 1000 mg vancomycin, 80 mg gentamicin and 1000 mg cefazolin in a 500 mL isotonic saline solution. The solution will be used to wash the dissected implant pocket and the implant prior to insertion in the implant pocket.
  Other Names: Hexamycin, Cefazolin "MIP" and Bactocin
  Arms: Irrigation of implants with a triple antibiotic solution
Other: Placebo — 500 mL of sterile isotonic (9%) saline. The solution will be used to wash the dissected implant pocket and the implant prior to insertion in the implant pocket.
  Other Names: Natriumklorid Fresenius Kabi 9 mg-ml
  Arms: Irrigation of implants with sterile isotonic saline

SUMMARY:
The BREAST-AB Trial is a multi-center, randomized, double blind, placebo-controlled trial investigating the efficacy of local application of gentamicin, vancomycin and cefazolin in decreasing all-cause implant explantation after breast reconstruction.

DETAILED DESCRIPTION:
The BREAST-AB Trial will include women undergoing breast reconstruction with implants. The objective is to determine the efficacy of local antibiotics in decreasing all-cause implant explantation. Participants will be randomized to local application of placebo or gentamicin, vancomycin and cefazolin in a saline solution onto the implant and the dissected breast pocket. All patients undergoing unilateral breast reconstruction will be randomized to the trial drug or placebo in a ratio of 1:1. All patients undergoing bilateral reconstruction will be randomized to the trial treatment on one of their breasts and placebo to the contralateral breast. A total number of 1274 of breasts undergoing breast reconstruction will be included in the trial.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Biologically female
* Signed informed consent
* Scheduled for breast reconstruction with implants or expanders including:

  1. Immediate or delayed reconstructions
  2. Bilateral or unilateral reconstructions
  3. With or without simultaneous flap reconstruction

Exclusion Criteria:

* Pregnancy
* Breast feeding
* Known allergy towards Vancomycin, Gentamicin and Cefazolin
* Known anaphylactic reaction towards other beta-lactam antibiotics or aminoglycosides
* Known allergy towards neomycin
* Known impaired renal function with GFR < 60 mL/min
* Participation in investigational drug trials and projects concerning disinfecting agents in the breast implant cavity
* Myasthenia Gravis

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1003 (Estimated)
Dates: Start 2021-01-27 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
All-cause explantation of the breast implant after the breast reconstruction surgery | 180 days
  All-cause explantation will be defined as explantation and discarding of the implant. Replacement of an expander with a permanent implant and replacement of a permanent breast implant with a new permanent breast implant due to cosmetic revisions such as asymmetry, implant malposition, change of size or implant rotation will not be counted as an explantation.

SECONDARY OUTCOMES:
Time to explantation (days) | 180 days
  Time to explantation will be defined as the amount of days between the breast reconstruction and the implant explantation surgery.
Revision surgery with incision of the fibrous capsule after the breast reconstruction surgery (Y/N) | 180 days
  The breast reconstruction surgery will be defined as the surgery where they received the allocated treatment
Exchange of permanent implant to expander implant after the breast reconstruction surgery (Y/N) | 180 days
  The breast reconstruction surgery will be defined as the surgery where they received the allocated treatment
Surgical site infection that leads to antibiotic treatment after the breast reconstruction surgery | 180 days
  Surgical site infection will be defined according to the CDC classification of surgical site infetion leading to antibiotic treatment with oral or intravenous antibiotics administered after the surgery.
All-cause explantation of the breast implant within 1 year after the breast reconstruction surgery | 1 year
  All-cause explantation will be defined as explantation and discarding of the implant. Replacement of an expander with a permanent implant and replacement of a permanent breast implant with a new permanent breast implant due to cosmetic revisions such as asymmetry, implant malposition, change of size or implant rotation will not be counted as an explantation.

OTHER OUTCOMES:
Time from the breast reconstruction surgery to discharge (days) | 180 days
  Time to discharge will be defined as the amount of days between the breast reconstruction and the day of discharge.
Re-admission after the breast reconstruction surgery (Y/N) | 180 days
  The breast reconstruction surgery will be defined as the surgery where the patient received the allocated treatment.
Long term follow-up after 5, 10 and 15 years | 15 years
  Capsular contracture and the Baker classification grade will be obtained from the National Patient Registry and the patients' medical journals after 5, 10 and 15 years. The BREAST-Q questionnaire will be used to assess patient-reported outcomes. The patients will be contacted and asked to fill out the questionnaire with 5 year-intervals after the surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Mikkel Herly, MD, Ph.D., Principal Investigator — Department of Plastic Surgery and Burns Treatment
Locations (8):
- Denmark (8):
  - Aalborg University Hospital, Aalborg
  - Aarhus University Hospital, Aarhus
  - Rigshospitalet, Copenhagen
  - South-West Jutland Hospital, Esbjerg
  - Herlev and Gentofte Hospital, Herlev
  - Odense University Hospital, Odense
  - Zealand University Hospital, Roskilde
  - Vejle Hospital, Vejle

IPD SHARING:
Plan to Share IPD: Yes
The protocol including the statistical analysis plan is published in BMJ Open (doi:10.1136/bmjopen-2021-058697) prior to unblinding. The main article will include the primary and secondary outcomes. The tertiary and long-term outcomes will be included in subsequent articles. The manuscripts will be submitted to peer-reviewed international journals and both positive, negative and inconclusive results will be published. The findings of the trial will be shared with participating sites and presented at national and international conferences. The results will be disseminated to the public but will not be shared directly with participating patients.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After the end of the trial, the data will become available (Anticipated july 2025)
Access Criteria: Researchers and other relevant parties can be granted access to selected anonymized data after publication upon request to the principal-sponsor investigator

REFERENCES:
- [Derived] Hemmingsen MN, Larsen A, Weltz TK, Orholt M, Wiberg S, Bennedsen AK, Bille C, Carstensen LF, Jensen LT, Bredgaard R, Koudahl V, Schmidt VJ, Vester-Glowinski P, Holmich LR, Sorensen SJ, Bjarnsholt T, Damsgaard T, Herly M. Prophylactic treatment of breast implants with a solution of gentamicin, vancomycin and cefazolin antibiotics for women undergoing breast reconstructive surgery: protocol for a randomised, double-blind, placebo-controlled trial (The BREAST-AB trial). BMJ Open. 2022 Sep 17;12(9):e058697. doi: 10.1136/bmjopen-2021-058697. PMID 36115667
- See also: Study protocol published in BMJ Open — https://bmjopen.bmj.com/content/12/9/e058697.abstract

DOCUMENTS (2):
  • Study Protocol: Study protocol v3.0 20/11/2025 incl. cover page (2025-11-20): https://cdn.clinicaltrials.gov/large-docs/25/NCT04731025/Prot_002.pdf
  • Statistical Analysis Plan: Statistical analysis plan v1.0 30/01/2026 incl. cover page (2026-01-30): https://cdn.clinicaltrials.gov/large-docs/25/NCT04731025/SAP_003.pdf